CLINICAL TRIAL: NCT01744925
Title: An Open-label,Randomized,Controlled Study to Evaluate the Safety and Efficacy for Icotinib at Different Doses in Second-line Treatment for Non-small Cell Lung Cancer Patients With Wild Type EGFR
Brief Title: Icotinib at Different Doses in Second-line Treatment for Non-small Cell Lung Cancer Patients With Wild Type EGFR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV26
Record Dates: First submitted 2012-12-05; First posted 2012-12-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2012-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Icotinib of routine dose (Active Comparator): Icotinib: 125mg, oral administration, three times per day.
  Interventions: Drug: Icotinib of routine dose
- Icotinib of high dose (Experimental): Icotinib: 375mg, oral administration, three times per day.
  Interventions: Drug: Icotinib of high dose

INTERVENTIONS:
Drug: Icotinib of routine dose — Icotinib: 125mg, oral administration, three times per day.
  Other Names: Conmana; BPI-2009
  Arms: Icotinib of routine dose
Drug: Icotinib of high dose — Icotinib: 375mg, oral administration, three times per day.
  Other Names: BPI-2009; Conmana
  Arms: Icotinib of high dose

SUMMARY:
This study is designed to evaluate the safety and efficacy of icotinib at routine dose and higher dose as second-line treatment in non-small cell lung cancer patients with epidermal growth factor receptor of wild type.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or progressive Non-Small Cell Lung Cancer stage IV or IIIB patients with Histologic or cytologic confirmation.
* Wild type epidermal growth factor receptor status.
* Progressed after first-line chemotherapy.
* No previous systemic anticancer therapy.
* Measurable lesion according to response evaluation criteria in solid tumors with at least one measurable lesion not previously irradiated.
* Provision of written informed consent.

Exclusion Criteria:

* Evidence of clinically active Interstitial Lung Diseases (Patients with chronic, stable, radiographic changes who are asymptomatic need not be excluded).
* Positive epidermal growth factor receptor mutation.
* Known severe hypersensitivity to icotinib or any of the excipients of this product.
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 4 weeks
  Number of participants with an objective response. An objective response (OR) was defined as a patient having a best overall response of either complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors, confirmed at least 28 days following the date of the initial response.

SECONDARY OUTCOMES:
Progression free survival | 3 months
  Progression free survival was defined as the time from the date of first dose of study medication to the date of first documentation of tumor progression or death due to any cause, whichever occurred first.
Overall survival | 14 months
  Overall Survival was assessed via calculation of the time to death due to any cause. If a participant was known to have died, the time to death was defined as the time from the date of randomization to the date of death. Otherwise, a participant was censored at the last date they were known to be alive.
Number of Participants with Adverse Events | 18 months
  Adverse events, Serious adverse events , incidence of and reason for study drug dose interruptions and discontinuations, laboratory assessments, vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Changli Wang, M.D., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China